CLINICAL TRIAL: NCT05100797
Title: Validity of the Vyntus CPX Metabolic Cart for Assessing Postprandial Energy Expenditure and Respiratory Exchange Ratio
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Principal Investigator, Universidad de Granada
Other Study IDs: 2190/CEIH/2021
Record Dates: First submitted 2021-09-16; First posted 2021-10-29 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vyntus CPX — To study the validity, precision and accuracy of the Vyntus CPX metabolic cart using both, in-vitro and in-vivo (i.e., human study) measures.

SUMMARY:
The aims of the present study are described below:

Aim 1: In-vitro measures to determine the validity, precision and accuracy of the Vyntus CPX metabolic cart assessed by:

1.1. Methanol burning tests. 1.2. Pure gas (nitrogen [N2] and carbon dioxide [CO2]) infusions to simulate both, constant and variable fluxes of oxygen consumption (VO2) and carbon dioxide production (VCO2) in different conditions and moments.

1. Immediately after or prior the methanol burning test (in a randomized order).
2. In separate days and time-periods.

Aim 2: In-vivo measures using the Vyntus CPX metabolic cart:

2.1. To assess the resting metabolic rate (RMR or resting energy expenditure [REE]) and respiratory exchange ratio (RER) day-to-day biological reproducibility (i.e. reliability) of the metabolic cart.

2.2. Further, the investigators will use an oral glucose tolerance test (OGTT) to determine the post-prandial day-to-day biological reproducibility (especifically the post-prandial RER) of the metabolic cart.

DETAILED DESCRIPTION:
The study will be developed in three different experiments which are detailed below:

EXPERIMENT 1 (AIM 1.1 AND 1.2.A):

The investigators will determine the Vyntus CPX measurement error over 14 different days by using both, methanol burnings and pure gas infusions. The order will be random.

1. Methanol burning: the investigators will burn the methanol inside the glass-cage and the investigators will measure dynamically the weight of burned alcohol; gas exchange will be continuously measured with the Vyntus CPX while the produced gases are directed into the metabolic cart's hose tube. The burning will take approximately 25-30 minutes and is expected to produce a RER=0.667.
2. Pure gas infusions: Pure N2 (concentration ≥99.9997%) for diluting ambient O2 and CO2 (concentration ≥99.995%) will be infused using high-precision mass-flow controllers (358 Series, Analyt-MTC, Müllheim, Germany; 0-2 l/min) into the metabolic cart's hose tube. The infused volumes of N2 and CO2 will be selected to replicate (i.e. mimic) as much as possible the VO2 and VCO2 produced by the methanol burning test. The gas infusions will last 20 minutes.

EXPERIMENT 2 (AIM 1.2.B):

The investigators will determine the Vyntus CPX measurement error over 14 different days by using pure gas infusions (each pure gas infusion will last 20 minutes). The procedures will be as follow:

1. Pure gas infusions varying, in a random order, the simulated VO2 and VCO2 to poduce different energy expenditure (EE) and RER values: the investigators will infuse pure N2 and CO2 gases at different volumes. The infusions will be performed either in the morning or in the afternoon (i.e. random) in 14 different and separate days. The randomly selected simulated EE will range between 1000 and 2000 kilocalories per day (kcal/day) while the RER will range between 0.80 and 0.95. The investigators will perform 5 pure gas infusions per day.
2. Pure gas infusions varying, in a random order, the simulated VO2 and VCO2 to produce different EE values while keeping a constant RER: the investigators will infuse pure N2 and CO2 gases at different volumes. The infusions will be performed either in the morning or in the afternoon (i.e. random) in 14 different and separate days. The randomly selected simulated EE will range between 1000 and 2000 kcal/day while the RER is fixed at 0.85. The investigators will perform 5 pure gas infusions per day.
3. Pure gas infusions varying, in a random order, the simulated VO2 and VCO2 to produce different RER values while keeping a constant EE: the investigators will infuse pure N2 and CO2 gases at different volumes. The infusions will be performed either in the morning or in the afternoon (i.e. random) in 14 different and separate days. The randomly selected simulated RER will range between 0.80 and 0.95 while the EE is fixed at 1500 kcal/day. The investigators will perform 5 pure gas infusions per day.

EXPERIMENT 3 (AIM 2.1 and 2.2.):

The investigators will assess the RMR and RER of 10-15 young-healthy adults using the Vyntus CPX metabolic cart on two consecutive days in the morning. The assessment will last 30 minutes and will be performed in agreement with current guidelines. The subjects will lay on a reclined bed in supine position and covered by a bed sheet for 20 minutes before the assessment as an 'acclimation period'. Immediately after this acclimation period the RMR and RER assessment will start under the same conditions. Then, the glucose beverage (75g of glucose/200ml) is given to the participants and another 180 minutes of assessment are performed.

In addition, the participants' weight, height and body composition (using a dual X-ray absorptiometry scan [DXA scan]) will be measured upon arrival on the first visit. Blood samples will be collected at different time periods to determine the blood glucose concentration. Lastly, participants will be asked to consume a standardized dinner (specifically designed by a dietitians team) the night before each study day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy.
* Age 18-40 y.
* BMI between 18.5 kg/m2 and 30 kg/m2 (both inclusive).
* Willing to fast and not to consume non-caloric stimulant for 12h before the assessments.
* Willing to avoid moderate or vigorous physical activity during 24-48h respectively.
* Have a stable body weight over the last 3 months (changes ≤3 kg) and not being enrolled in a weight loss program.

Exclusion Criteria:

* Smoking or use of tobacco products within the last 3 months.
* Diagnosed with diabetes.
* Previous bariatric surgery (or other surgeries) for obesity or weight loss.
* Use of medications affecting metabolism or sleep.
* History of neurological disease.
* History of cardiovascular disease, including hypertension, or other chronic diseases.
* Pregnant, planning to become pregnant, or breastfeeding.
* Adherence to special restrained diets (e.g., low-carbohydrates, low-fat, or vegetarian/vegan diets) over the last 3 months.
* Claustrophobia impeding to stay calm under a plastic canopy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: To be included in the study, the participants have to be healthy and meet the abovementioned inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-02-23 (Estimated); Study Completion 2022-03-23 (Estimated)

PRIMARY OUTCOMES:
VO2 post-prandial gas exchange assessed by indirect calorimetry | 5 hours
  Volume of oxygen consumption (VO2 [ml/min])
VCO2 post-prandial gas exchange assessed by indirect calorimetry | 5 hours
  Volume of carbon dioxide production (VCO2 [ml/min])
EE post-prandial gas exchange assessed by indirect calorimetry | 5 hours
  -Energy Expenditure (EE [kcal/day])
RER post-prandial gas exchange assessed by indirect calorimetry | 5 hours
  Respiratory Exchange Ratio (RER [calculated as VCO2-to-VO2 ratio])
CHOox post-prandial gas exchange assessed by indirect calorimetry | 5 hours
  Carbohydrate oxidation (CHOox [g/min])
FATox post-prandial gas exchange assessed by indirect calorimetry | 5 hours
  Fat oxidation (FATox [g/min])
VO2 validity of the metabolic cart. In-vitro measurements and/or simulations to determine the validity, precision and accuracy of the metabolic cart assessed by methanol burning tests and controlled pure gas infusions. | 14 separate days; measurements of 2 hours per day
  Volume of oxygen consumption (VO2) measurement error (ml/min)
VCO2 validity of the metabolic cart. In-vitro measurements and/or simulations to determine the validity, precision and accuracy of the metabolic cart assessed by methanol burning tests and controlled pure gas infusions. | 14 separate days; measurements of 2 hours per day
  Volume of carbon dioxide production (VCO2) measurement error (ml/min)
EE validity of the metabolic cart. In-vitro measurements and/or simulations to determine the validity, precision and accuracy of the metabolic cart assessed by methanol burning tests and controlled pure gas infusions. | 14 separate days; measurements of 2 hours per day
  Energy Expenditure (EE) measurement error (kcal/day)
RER validity of the metabolic cart. In-vitro measurements and/or simulations to determine the validity, precision and accuracy of the metabolic cart assessed by methanol burning tests and controlled pure gas infusions. | 14 separate days; measurements of 2 hours per day
  Respiratory Exchange Ratio (RER) measurement error

SECONDARY OUTCOMES:
Post-prandial blood glucose concentrations | 5 hours
  Measures of blood glucose concentrations (mg/dl)
Body composition outcomes (DXA scann) | 1 day
  Lean mass, fat-free mass and fat mass in kilograms
Anthropometric measurements 1, weight | 1 day
  Weight in kilograms
Anthropometric measurements 2, height | 1 day
  Height in meters
Anthropometric measurements 3, body mass index | 1 day
  BMI: Weight and height will be combined to report in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No